CLINICAL TRIAL: NCT01896219
Title: Multicentric Evaluation of IMACTIS-CT Navigation System
Brief Title: CTNAV II : Multicentric Evaluation of IMACTIS-CT Navigation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 12 29; 2013-A00539-36 (Other: IDRCB)
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Drainage; Biopsy; Punction; Ablation
Keywords: Medical device; CT; Needle; Navigation; IMACTIS-CT®; Thoraco-abdominal level; anesthesia needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gesture performed under control tomodensitometric (CT) (Active Comparator): Conventional
  Interventions: Device: CT
- Gesture performed under Navigation-assisted procedure (NAV) (Experimental): Use of the IMACTIS-CT® Navigation System
  Interventions: Device: Navigation station (IMACTIS-CT®)

INTERVENTIONS:
Device: Navigation station (IMACTIS-CT®)
  Other Names: Navigation station for gestures (carried out under CT) guidance
  Arms: Gesture performed under Navigation-assisted procedure (NAV)
Device: CT — Reference method for gestures (carried out under CT) guidance
  Arms: Gesture performed under control tomodensitometric (CT)

SUMMARY:
Estimate the medical service of a system of navigation (IMACTIS-CT®)in terms of SAFETY, EFFICIENCY and PERFORMANCE, in comparison with the reference method during gestures of interventional radiology under scan in the thoraco-abdominal level.

ELIGIBILITY:
Inclusion Criteria:

* More or equal the 18 years old
* Patient for whom an indication of diagnostic or therapeutic percutaneous interventional gesture in the thoraco-abdominal level under CT guidance is prescribed
* Patient affiliated to social security or similarly regime
* Patient signed consent for participation in the study.

Exclusion Criteria:

* Patient with a medical device using a magnetic field (eg, patient with a pacemaker)
* Patient who presents ferromagnetic foreign bodies intracorporeal close to the working zone of Radiologist, and that can interact with the medical device
* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Person deprived of freedom by judicial or administrative decision
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Estimate the medical service of a system of navigation (IMACTIS-CT ®) in terms of SAFETY, EFFICIENCY and PERFORMANCE, in comparison with the reference method during interventional radiology gestures | 2 hours
  Three criteria are estimated:
  * Safety: number of major complications (due to gesture)
  * Efficiency: number of targets achieved
  * Performance: number of scancontrol made during the puncture

SECONDARY OUTCOMES:
Comparison of the duration of needle setting up procedure between IMACTIS-CT® and the reference method. | 2 hours
Comparison (IMACTIS-CT ® vs References) of the operator satisfaction during his gesture. | 2 hours
  Scale of quantitative satisfaction
Comparison (IMACTIS-CT ® vs. Reference) of the radiation dose delivered during the puncture. | 2 hours
Evaluation of delivered medical service by carrying out a sub-group analysis according to the stratification of the difficulty of gesture | 2 hours
Evaluation of the navigation system use by the operators, based on needle holder localization files | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bricault, Pr, Principal Investigator — Radiology Departement - University Hospital of Grenoble; Eric Delabrousse, Pr, Principal Investigator — University Hospital of Besançon; Bruno Lapuyade, MD, Principal Investigator — University Hospital, Bordeaux; Pascal Lacombe, Pr, Principal Investigator — University Hospital of Garches; Laurent Lemaitre, Pr, Principal Investigator — University Hospital of Lille; Valérie Laurent, Pr, Principal Investigator — CHU NANCY; Jean-Yves Gauvrit, Pr, Principal Investigator — University Hospital of Rennes; Olivier Favelle, MD, Principal Investigator — University Hospital of Tours; Eric De Kerviler, Pr, Principal Investigator — University Hospital of Saint-Louis
Locations (9):
- France (9):
  - University Hospital, Besançon, Doubs
  - University Hospital, Bordeaux, Gironde
  - Ambroise Paré University Hospital, Boulogne-Billancourt, Hauts-de-Seine
  - University Hospital, Rennes, Ille-et-Vilaine
  - University Hospital, Tours, Indre-et-Loire
  - University Hospital, Grenoble, Isère
  - University Hospital, Nancy, Meuse
  - University Hospital, Lille, Nord
  - University Hospital of Saint-Louis, Paris

REFERENCES:
- [Derived] Rouchy RC, Moreau-Gaudry A, Chipon E, Aubry S, Pazart L, Lapuyade B, Durand M, Hajjam M, Pottier S, Renard B, Logier R, Orry X, Cherifi A, Quehen E, Kervio G, Favelle O, Patat F, De Kerviler E, Hughes C, Medici M, Ghelfi J, Mounier A, Bricault I. Evaluation of the clinical benefit of an electromagnetic navigation system for CT-guided interventional radiology procedures in the thoraco-abdominal region compared with conventional CT guidance (CTNAV II): study protocol for a randomised controlled trial. Trials. 2017 Jul 6;18(1):306. doi: 10.1186/s13063-017-2049-6. PMID 28683837